CLINICAL TRIAL: NCT01618305
Title: A Phase IV Randomized Trial to Evaluate the Virologic Response and Pharmacokinetics of Two Different Potent Regimens in HIV Infected Women Initiating Triple Antiretroviral Regimens Between 20 and 36 Weeks of Pregnancy for the Prevention of Mother-to-Child Transmission: NICHD P1081
Brief Title: Evaluating the Response to Two Antiretroviral Medication Regimens in HIV-Infected Pregnant Women, Who Begin Antiretroviral Therapy Between 20 and 36 Weeks of Pregnancy, for the Prevention of Mother-to-Child Transmission
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Westat (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: P1081; 10770 (Registry Identifier: DAIDS ES Registry Number); NICHD P1081; HHSN2752018000011. (Other Grant/Funding Number: NICHD); UM1AI068616 (NIH)
Record Dates: First submitted 2012-06-06; First posted 2012-06-13 (Estimated); Results first posted 2019-12-26 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — lamivudine, zidovudine drug combination; efavirenz; Raltegravir Potassium

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Arm A (Women) (Experimental): Pregnant women received ZDV/3TC + EFV
  Interventions: Drug: Lamivudine/zidovudine; Drug: Efavirenz
- Arm B (Women) (Experimental): Pregnant women received ZDV/3TC + RAL
  Interventions: Drug: Lamivudine/zidovudine; Drug: Raltegravir
- Arm A (Infants) (No Intervention): Infants born to women in Arm A; infants received no study intervention.
- Arm B (Infants) (No Intervention): Infants born to women in Arm B; infants received no study intervention.

INTERVENTIONS:
Drug: Lamivudine/zidovudine — Participants received one lamivudine 150 mg/zidovudine 300 mg fixed-dose combination tablet twice a day from entry through delivery*.
  * Participants may have received a locally supplied nucleoside reverse transcriptase inhibitor (NRTI) backbone in place of lamivudine/zidovudine with permission of the protocol team obtained prior to randomization.
  Other Names: ZDV/3TC
  Arms: Arm A (Women); Arm B (Women)
Drug: Efavirenz — Participants received one 600 mg tablet of efavirenz each night from entry through delivery.
  Other Names: EFV
  Arms: Arm A (Women)
Drug: Raltegravir — Participants received one 400 mg raltegravir tablet twice a day from entry through delivery.
  Other Names: RAL
  Arms: Arm B (Women)

SUMMARY:
HIV-infected pregnant women who begin taking antiretroviral (ARV) medications in the late stages of pregnancy need an effective medication regimen to reduce the risk of transmitting HIV to their children. This study examined the virologic response, safety, and tolerability of two different ARV medication regimens in HIV-infected pregnant women who were between 20 and 36 weeks pregnant when they entered the study.

DETAILED DESCRIPTION:
When initiating this study there were many ARV medications and combination regimens available to treat HIV-infected people. However, the number of ARV medications that had been studied in HIV-infected pregnant women for the prevention of mother-to-child transmission was limited. Although HIV-infected pregnant women who began taking ARV medications late in their pregnancies required effective therapy to reduce the risk of transmitting HIV to their children, there were no published data available that compared the effects of non-nucleoside reverse transcriptase inhibitors (NNRTI) and integrase inhibitors (which are two classes of ARV medications) in pregnant women. The purpose of this study was to compare the safety, tolerability, and virologic responses to two different medication regimens, each of which included an NNRTI or integrase inhibitor, in pregnant HIV-infected women who began ARV therapy late in their pregnancies (i.e., had gestational age between 20 and 36 weeks).

This study was originally opened under IMPAACT P1081, protocol version 2.0 (version 1.0 never opened to accrual) as a three arm study. However, IMPAACT P1081 was closed due to slow accrual, at which point NICHD took over the study, streamlined it to two arms, and reopened it as NICHD P1081 under protocol Version 3.0. Women who enrolled under IMPAACT P1081 (N=20) and were randomized to one of the two continuing arms (efavirenz- or raltegravir-based ART; N=14) were included in NICHD P1081, while IMPAACT P1081 women randomized to the dropped arm (lopinavir/ritonavir-based ART; N=6) were not eligible for inclusion in NICHD P1081.

In this study HIV-infected pregnant women were randomly assigned to one of two arms. Women in Arm A received lamivudine 150 mg/zidovudine 300 mg twice a day and efavirenz 600 mg each night. Women in Arm B received lamivudine 150 mg/zidovudine 300 mg twice a day and raltegravir 400 mg twice a day. All women were scheduled to receive their assigned medications from study entry through delivery. Antepartum study visits were scheduled at entry and Weeks 1, 2, and 4; and thereafter, every two weeks until labor and delivery. Study visits included a medical history review, physical examination, questionnaires, blood collection, and a vaginal swab procedure.

While women were in labor, they were scheduled to continue to receive their study medications. Some women may have received additional or alternate medications according to local standard of care/guidelines. Women had a physical examination and blood collection at the delivery visit. After delivery, some women continued to receive ARV medications according to the local guidelines, and could have received study ARV for up to eight weeks postpartum while they transitioned to the ARV regimen indicated per their local standard of care. Women were scheduled to attend study visits following delivery at Weeks 2, 6, 16, and 24, which included a medical history review, physical examination, and blood collection. Select visits were scheduled to include a vaginal swab procedure. Some women had vaginal specimens stored for future research.

Infants delivered on study were scheduled to receive ARV medications as prescribed by the babies' doctors per local standard of care/guidelines. Study visits for infants were scheduled at birth, and at Weeks 2, 6, 16, and 24. Each study visit included a medical history review, physical examination, and blood collection. Select visits included oral and nasopharyngeal swab collection.Some infants had oral and/or nasopharyngeal specimens stored for future research.

ELIGIBILITY:
Inclusion Criteria:

* Naive to antiretroviral therapy (ART) or have received ART with short course zidovudine (maximum of 8 weeks) for prevention of mother-to-child transmission in previous pregnancies
* Willing and able to sign informed consent. Participant must be of an age to provide legal informed consent as defined by the country in which the participant resides. If not, the informed consent must be signed by a legal guardian/parent, as per country guidelines.
* Documentation of HIV-1 infection defined as positive results from two samples collected at different time points. The same method may be used at both time points. All samples tested must be whole blood, serum, or plasma. Documentation may be abstracted from medical records to satisfy these criteria for infection. More information on this criterion can be found in the protocol.
* Viable pregnancy with gestational age of greater than or equal to 20 weeks to less than or equal to 36 weeks based upon menstrual history and/or ultrasound. Note: If menstrual history is unknown or if there is a discrepancy between menstrual history and ultrasound, determination of gestational age should be based upon best available methodology at each site.
* Intends to continue pregnancy
* Willingness and intent to deliver at the participating clinical site and to be followed for the duration of the study at the site or associated outpatient facility
* Willing to comply with the study regimen
* Agrees to use two reliable methods of contraception after delivery if randomized to the efavirenz arm and is sexually active. A barrier method of contraception (condoms, diaphragm, or cervical cap) together with another reliable form of contraception must be used for 4 weeks after stopping efavirenz.

Exclusion Criteria:

* Active labor defined as onset of regular contractions or cervical dilatation greater than 2 cm
* Use of ART during current pregnancy
* Chemotherapy for active malignancy
* HIV genotypic resistance, as defined in the protocol, to efavirenz or raltegravir or to NRTIs that will be included in the ART regimen. Note: A lack of HIV drug resistance test results at the time of enrollment is not exclusionary.
* Serious active opportunistic infection and/or serious bacterial infection including active tuberculosis (TB) or unstable or severe medical condition within 14 days of study entry
* Active drug or alcohol use or dependence that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Any clinically significant diseases (other than HIV infection) or clinically significant findings during the screening medical history or physical examination that, in the investigator's opinion, would compromise the outcome of this study
* Vomiting or inability to swallow medications due to an active, pre-existing condition that prevents adequate swallowing and absorption of study medication
* Known allergy/sensitivity to any study drugs or their formulations or sulfonamide allergy
* The following laboratory values (within 30 days of enrollment):

  1. Hemoglobin greater than or equal to Grade 3
  2. Absolute neutrophil count greater than or equal to Grade 2
  3. Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) greater than or equal to Grade 2
  4. Serum creatinine greater than or equal to Grade 1
  5. Platelet count greater than or equal to Grade 3
* Evidence of pre-eclampsia (such as persistent diastolic blood pressure greater than 90 mm Hg)
* Receipt of disallowed medications as described in the protocol

Min Age: 16 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2013-09-05 (Actual); Primary Completion 2018-12-11 (Actual); Study Completion 2018-12-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Esau Joao, M.D., Study Chair — Hospital Federal dos Servidores do Estado - RJ; Mark Mirochnick, M.D., Study Chair — Boston Medical Center
Locations (19):
- United States (4):
  - South Flordia Childrens Diagnostic & Treatment Center, Fort Lauderdale, Florida
  - Tulane University, New Orleans, Louisiana
  - St Jude's Children's Research Hospital, Memphis, Tennessee
  - University of Washington Medical Center, Seattle, Washington
- Argentina (2):
  - Hosp. General de Agudos Buenos Aires Argentina NICHD CRS, Ciudad de Buenos Aires, Buenos Aires
  - Fundacion Huesped - Hospital Juan A Fernandez, Buenos Aires
- Brazil (7):
  - SOM Federal University Minas Gerais Brazil NICHD CRS, Belo Horizonte, Minas Gerais
  - Univ. Caxias do Sul Brazil NICHD CRS, Caxias do Sul, Rio Grande do Sul
  - Hospital Nossa Senhora da Conceicao NICHD CRS, Porto Alegre, Rio Grande do Sul
  - Hospital Federal dos Servidores do Estado NICHD CRS, Rio de Janeiro
  - Instituto de Puericultura e Pediatria Martagao Gesteira - UFRJ NICHD CRS, Rio de Janeiro
  - Hosp. Geral De Nova Igaucu Brazil NICHD CRS, Rio de Janeiro
  - Univ. of Sao Paulo Brazil NICHD CRS, São Paulo
- San Juan City Hosp. PR NICHD CRS, San Juan, Puerto Rico
- Perinatal HIV Research Unit-Chris Hani Baragwanath Hospital, Soweto, South Africa
- Kilimanjaro Christian Medical Centre (KCMC), Moshi, Tanzania
- Thailand (3):
  - Siriraj Hospital ,Mahidol University NICHD CRS, Bangkok, Bangkoknoi
  - Bhumibol Adulyadej Hospital, Bangkok
  - Chiangrai Prachanukroh Hospital NICHD CRS, Chiang Mai

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie results in the publication, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: Beginning 9 months following publication and available throughout period of funding of the Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) by NIH.
Access Criteria: With whom? Researchers whose proposed use of the data is approved by the NICHD Data and Specimen Hub (DASH) Data Access Committee as scientifically and ethically appropriate and does not conflict with constraints or informed consent limitations.
  For what types of analyses? To achieve aims in the approved proposal. By what mechanism will data be made available? To gain access, data requestors will need to create a free NICHD DASH account, submit a data access proposal, and if approved, sign a data access agreement. Information regarding creating a NICHD DASH account and accessing data may be found at https://dash.nichd.nih.gov/

REFERENCES:
- [Derived] Joao EC, Morrison RL, Shapiro DE, Chakhtoura N, Gouvea MIS, de Lourdes B Teixeira M, Fuller TL, Mmbaga BT, Ngocho JS, Njau BN, Violari A, Mathiba R, Essack Z, Pilotto JHS, Moreira LF, Rolon MJ, Cahn P, Prommas S, Cressey TR, Chokephaibulkit K, Werarak P, Laimon L, Hennessy R, Frenkel LM, Anthony P, Best BM, Siberry GK, Mirochnick M. Raltegravir versus efavirenz in antiretroviral-naive pregnant women living with HIV (NICHD P1081): an open-label, randomised, controlled, phase 4 trial. Lancet HIV. 2020 May;7(5):e322-e331. doi: 10.1016/S2352-3018(20)30038-2. PMID 32386720
- See also: The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 2.0, November 2014 (Corrected to Version 2.1, July 2017). — https://rsc.niaid.nih.gov/clinical-research-sites/daids-adverse-event-grading-tables
- See also: The Division of AIDS Manual for the Expedited Reporting of Adverse Events, Version 2.0, January 2010. — https://rsc.niaid.nih.gov/clinical-research-sites/manual-expedited-reporting-adverse-events-daids

RESULTS

PARTICIPANT FLOW:
Recruitment Details: IMPAACT P1081 (protocol version 2.0) enrolled participants from September, 2013 through November, 2014. Enrollment under NICHD P1081 (protocol version 3.0) resumed in July 2015 and continued through February, 2018. Participants enrolled at sites in Argentina (2), Brazil (7), South Africa (1), Tanzania (1), Thailand (3), and the United States (5).
Pre-assignment Details: Participants were randomized 1-to-1 to Arm A (efavirenz) or Arm B (raltegravir) with stratification by gestational age at enrollment (20 to <28 weeks; 28 to <31 weeks; 31 to <34 weeks; 34 to <37 weeks) and NRTI backbone (lamivudine/zidovudine or alternative, locally-supplied NRTI regimen), and dynamic balancing by study site.
Groups:
- Arm A (Women): Pregnant women received ZDV/3TC + EFV
  Lamivudine/zidovudine: Participants received one lamivudine 150 mg/zidovudine 300 mg fixed-dose combination tablet twice a day from entry through delivery*.
  * Participants may have received a locally supplied nucleoside reverse transcriptase inhibitor (NRTI) backbone in place of lamivudine/zidovudine with permission of the protocol team obtained prior to randomization.
  Efavirenz: Participants received one 600 mg tablet of efavirenz each night from entry through delivery.
- Arm B (Women): Pregnant women received ZDV/3TC + RAL
  Lamivudine/zidovudine: Participants received one lamivudine 150 mg/zidovudine 300 mg fixed-dose combination tablet twice a day from entry through delivery*.
  * Participants may have received a locally supplied nucleoside reverse transcriptase inhibitor (NRTI) backbone in place of lamivudine/zidovudine with permission of the protocol team obtained prior to randomization.
  Raltegravir: Participants received one 400 mg raltegravir tablet twice a day from entry through delivery.
Period: Overall Study
Arm/Group | Arm A (Women) | Arm B (Women)
Started | 202 | 206
Completed | 187 | 196
Not Completed | 15 | 10
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 11 | 7
Not completed — Protocol Violation | 1 | 0
Not completed — Withdrawal by Subject | 3 | 2

BASELINE CHARACTERISTICS:
Population: All women randomized to NICHD P1081 were eligible for inclusion in this summary. Additionally, the 14 women who were randomized under IMPAACT P1081 to one of the two continuing arms in NICHD P1081 were also eligible for inclusion.
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A (Women) | Arm B (Women) | Total
Number analyzed (Participants) | 202 | 206 | 408
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 25.4 [21.8 to 31.0] | 26.9 [22.6 to 31.8] | 26.5 [22.2 to 31.5]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 202 | 206 | 408
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian, Pacific Islander | 24 | 23 | 47
  Black, Not Hispanic | 74 | 72 | 146
  Hispanic, Latino | 101 | 108 | 209
  White, Not Hispanic | 1 | 2 | 3
  Unknown | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  Argentina | 8 | 12 | 20
  Puerto Rico | 0 | 2 | 2
  United States | 4 | 1 | 5
  Tanzania | 42 | 42 | 84
  Brazil | 94 | 96 | 190
  South Africa | 30 | 30 | 60
  Thailand | 24 | 23 | 47
HIV-1 RNA Plasma Viral Load [Median (Inter-Quartile Range); unit: Log10 copies/mL] — Population: Five women (two in the Arm A and three in Arm B) were missing HIV-1 RNA viral load at entry.
  Log10 copies/mL
    number analyzed (Participants) | 200 | 203 | 403
    (all) | 4.1 [3.4 to 4.5] | 4.1 [3.3 to 4.6] | 4.1 [3.4 to 4.6]
Absolute CD4 Count [Median (Inter-Quartile Range); unit: cells/mm^3] — Population: Eleven women (seven in Arm A and four in Arm B) were missing absolute CD4 cell count at baseline.
  cells/mm^3
    number analyzed (Participants) | 195 | 202 | 397
    (all) | 408 [289 to 602] | 389.5 [240 to 567] | 395 [262 to 574]
NRTI Background Regimen [Count of Participants; unit: Participants]
  Zidovudine and Lamivudine (ZDV/3TC) | 170 | 171 | 341
  Emtricitabine and Tenofovir (FTC/TDF) | 31 | 33 | 64
  Lamivudine and Tenofovir (3TC/TDF) | 1 | 2 | 3
Gestational Age [Count of Participants; unit: Participants]
  20-<28 weeks | 102 | 103 | 205
  28-<31 weeks | 48 | 50 | 98
  31-<34 weeks | 31 | 29 | 60
  34-<37 weeks | 21 | 24 | 45

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Women With Plasma HIV-1 RNA Viral Load Less Than 200 Copies/mL at Delivery
Description: If there was no viral load measurement at the delivery visit, the last viral load within three weeks prior to delivery was considered.
Time Frame: Measured at participants' delivery visit (or last visit within three weeks prior to delivery)
Population: Eligible women were those with plasma HIV-1 RNA viral load at (or within three weeks prior to) delivery. Evaluable women had HIV-1 RNA plasma viral load greater than or equal to 200 at entry (i.e. did not already have the outcome) and had resistance testing results (on a sample taken at screening) showing no genotypic resistance to any study drug.
Measure: Number; unit: Proportion
Arm/Group | Arm A (Women) | Arm B (Women)
Number analyzed (Participants) | 154 | 153
Proportion | .84 | .94
Statistical Analysis 1: Comparison: Arm A (Women) vs Arm B (Women); Test type: Superiority — P-value was calculated using a Cochran-Mantel-Haenszel test, stratified by gestational age at entry (20-<28 weeks; 28-<31 weeks; 31-<34 weeks; 34-<37 weeks); p = 0.001, Cochran-Mantel-Haenszel

2. Primary Outcome: Proportion of Participants Who Discontinued Randomized Study Drug Prior to Labor and Delivery.
Description: Only women who initiated (i.e. received at least one dose of) their randomized treatment were eligible for this outcome measure. Women were considered to have discontinued study drug if they stopped receiving efavirenz or raltegravir (whichever was assigned) prior to labor and delivery for any reason, including loss to follow-up.
Time Frame: Measured from entry through participants' delivery visit (approximately 36 to 40 weeks gestation)
Population: Five women (all in Arm A) never initiated treatment, and thus were not included in this outcome measure.
Measure: Number; unit: Proportion
Arm/Group | Arm A (Women) | Arm B (Women)
Number analyzed (Participants) | 197 | 206
Proportion | .05 | .03
Statistical Analysis 1: Comparison: Arm A (Women) vs Arm B (Women); Test type: Superiority; p = 0.557, Cochran-Mantel-Haenszel; The Cochran-Mantel-Haenszel test was stratified by gestational age at entry (20-<28 weeks; 28-<31 weeks; 31-<34 weeks; 34-<37 weeks)

3. Primary Outcome: Proportion of Women Who Experienced at Least One New Adverse Event of Greater Than or Equal to Grade 3 as Defined in the Division of AIDS (DAIDS) Toxicity Table
Description: "New" adverse events were those with an onset date on or after randomization. Adverse events present at baseline would only be considered "New" if they increased in grade on or after randomization.
  All women who received at least one dose of study drug were eligible for this analysis.
Time Frame: Measured from entry through participants' last study visit, approximately 24 weeks after delivery
Population: Five women (all in Arm A) never initiated their assigned study treatment and were not included in this analysis.
Measure: Number; unit: Propotion
Arm/Group | Arm A (Women) | Arm B (Women)
Number analyzed (Participants) | 197 | 206
Propotion | .30 | .30
Statistical Analysis 1: Comparison: Arm A (Women) vs Arm B (Women); Test type: Superiority; p = 0.909, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]

4. Primary Outcome: Proportion of Infants Who Experienced at Least One Adverse Event of Greater Than or Equal to Grade 3.
Description: All infants who were live births on study were eligible for this analysis. Adverse event grades were defined based on the DAIDS toxicity table.
Time Frame: Measured from birth through infants' last study visit, approximately 24 weeks after delivery
Population: All live born infants were included in this analysis.
Measure: Number; unit: Proportion
Arm/Group | Arm A (Infants) | Arm B (Infants)
Number analyzed (Participants) | 194 | 199
Proportion | .25 | .25
Statistical Analysis 1: Comparison: Arm A (Infants) vs Arm B (Infants); Test type: Superiority; p = 0.938, Cochran-Mantel-Haenszel; The Cochran-Mantel-Haenszel test was stratified by maternal gestational age at entry (20-<28 weeks; 28-<31 weeks; 31-<34 weeks; 34-<37 weeks)

5. Secondary Outcome: Proportion of Women Who Achieved HIV-1 RNA Virologic Suppression Below the Lower Limit of Quantification of the Assay at Delivery
Description: A successful outcome was defined as maternal HIV-1 RNA plasma viral load less than the lower limit of quantification (LLQ) for the testing assay, which could vary. Most (99%) women had their viral load measured using an assay with LLQ equal to 40 or 20 copies/mL.
  If the viral load at delivery was missing, the last observed viral load within 21 days prior to the delivery date was considered.
Time Frame: Measured at participants' delivery visit (or last visit within three weeks prior to delivery)
Population: Eligible women were those that had a plasma HIV-1 RNA viral load at (or within 21 days prior to) delivery. Evaluable women were those with HIV-1 RNA viral load >200 copies/mL at baseline, and results from genotypic testing performed on a sample taken at screening indicating no genotypic resistance to any study drug.
Measure: Number; unit: Proportion
Arm/Group | Arm A (Women) | Arm B (Women)
Number analyzed (Participants) | 154 | 153
Proportion | .58 | .86
Statistical Analysis 1: Comparison: Arm A (Women) vs Arm B (Women); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]

6. Secondary Outcome: Proportion of Women With 1) Successful Viral Load (Plasma HIV-1 RNA VL) Decrease From Entry to Week 2 and VL Less Than 1,000 Copies/ml at All Time Points After 4 Weeks on Study Drugs, Until Delivery; and 2) Who Remain on the Assigned Study Regimen
Description: A successful viral load decrease was defined as follows: for women having HIV-1 RNA viral load greater than or equal to 10,000 copies/mL at entry, a viral load <200 copies/mL; for women with VL less than 10,000 copies/mL at entry, a Log10 viral load decrease of at least 2.0 from entry.
Time Frame: Measured from entry through delivery (approximately 36 to 40 weeks gestation).
Population: Women were evaluable for this outcome measure if they had (1) a valid viral load result at Week 2 (day 11-17 after initiation of study drug), (2) initiated study drug, and (3) delivered on- study; evaluable women who delivered after 28 days on study drug additionally had (4) at least one viral load result after 28 days on study drug.
Measure: Number; unit: Proportion
Arm/Group | Arm A (Women) | Arm B (Women)
Number analyzed (Participants) | 133 | 139
Proportion | .63 | .89
Statistical Analysis 1: Comparison: Arm A (Women) vs Arm B (Women); Test type: Superiority; p < 0.001, Cochran-Mantel-Haenszel; [statistical method as in outcome 2, analysis 1]

7. Secondary Outcome: Log10 Change in Viral Load From Entry to Each Time Point Prior to Delivery
Description: Change in viral load from entry (or screening, if there was no entry viral load) to each study week prior to delivery, calculated on the log10 scale as log10(week X RNA) - log10(baseline RNA).
  For this analysis, HIV-1 RNA values that were censored below the lower limit of quantification (LLQ) were imputed to be equal to the LLQ - 1.
Time Frame: Measured at antepartum Weeks 1, 2, 4, 6, 8, 10, 12, 14, and 16.
Population: Women were included in each week below if they had not delivered prior to that week and had an RNA viral load result for that antepartum visit.
Measure: Median (Inter-Quartile Range); unit: Log10 copies/mL
Arm/Group | Arm A (Women) | Arm B (Women)
Number analyzed (Participants) | 183 | 185
Log10 copies/mL
  Week 1: number analyzed (Participants) | 179 | 185
  Week 1 | -1.4 [-1.7 to -1.2] | -1.5 [-1.8 to -1.2]
  Week 2: number analyzed (Participants) | 183 | 182
  Week 2 | -1.8 [-2.0 to -1.4] | -2.1 [-2.4 to -1.6]
  Week 4: number analyzed (Participants) | 175 | 176
  Week 4 | -2.0 [-2.3 to -1.6] | -2.4 [-2.8 to -1.6]
  Week 6: number analyzed (Participants) | 142 | 151
  Week 6 | -2.1 [-2.5 to -1.7] | -2.4 [-3.0 to -1.7]
  Week 8: number analyzed (Participants) | 133 | 133
  Week 8 | -2.2 [-2.6 to -1.7] | -2.4 [-3.0 to -1.7]
  Week 10: number analyzed (Participants) | 109 | 108
  Week 10 | -2.3 [-2.7 to -1.8] | -2.3 [-3.0 to -1.7]
  Week 12: number analyzed (Participants) | 82 | 99
  Week 12 | -2.4 [-2.7 to -1.9] | -2.5 [-3.0 to -1.8]
  Week 14: number analyzed (Participants) | 60 | 65
  Week 14 | -2.5 [-2.6 to -1.9] | -2.5 [-3.0 to -1.8]
  Week 16: number analyzed (Participants) | 49 | 45
  Week 16 | -2.5 [-2.7 to -1.8] | -2.7 [-3.0 to -2.1]

8. Secondary Outcome: Proportion of Women With HIV-1 RNA Plasma Viral Load Less Than 200 Copies/mL at Weeks 4 and 6 From Treatment Initiation
Description: The Week 4 and 6 participant viral loads were the viral load results obtained closest to (within four days of) the target date for that visit from initiation of treatment (for Week 4, day 24-32 after first dose; for Week 6, day 38-46 after first dose).
Time Frame: Measured at Weeks 4 and 6 from first dose of randomized treatment, prior to delivery
Population: Women were evaluable for Week 4 and/or Week 6 if they did not deliver prior to that study week and had at least one HIV-1 RNA plasma viral load obtained within 4 days of the target date from treatment initiation
Measure: Number; unit: Proportion
Arm/Group | Arm A (Women) | Arm B (Women)
Number analyzed (Participants) | 170 | 176
Proportion
  Week 4 | .75 | .95
  Week 6: number analyzed (Participants) | 140 | 151
  Week 6 | .85 | .96

9. Secondary Outcome: Proportion of Women With HIV-1 RNA Vaginal Viral Load Less Than 1200 Copies/mL at Weeks 4 and 6 From Treatment Initiation
Description: The Week 4 and 6 participant viral loads were the viral load results obtained closest to (within four days of) the target date for that visit from initiation of treatment (for Week 4, day 24-32 after first dose; for Week 6, day 38-46 after first dose).
  Vaginal swabs produce much less testable sample volume than blood plasma draws. Each vaginal swab specimen had to be diluted, and this dilution factor raised the lower limit of quantification (LLQ). The most commonly observed LLQs were 300 and 1200. For consistency, the higher LLQ was considered the threshold for this outcome measure.
Time Frame: Measured at Weeks 4 and 6 from first dose of randomized treatment, prior to delivery
Population: Participants were included if they had a valid RNA results at Week 4 and/or Week 6, and had not delivered prior to obtaining the viral load measurement for that week.
Measure: Number; unit: Proportion
Arm/Group | Arm A (Women) | Arm B (Women)
Number analyzed (Participants) | 159 | 168
Proportion
  Week 4 | .97 | .95
  Week 6: number analyzed (Participants) | 137 | 143
  Week 6 | .98 | .94

10. Secondary Outcome: Infectivity of Plasma
Description: The goal of this outcome measure was to address an objective relevant to protease inhibitors, one of which was originally included as a third arm in the Version 2.0 of the study. This outcome measure was included to assess how the infectivity of plasma changed over time among women receiving protease inhibitors, and whether this differed from other classes of antiretroviral drugs. However, the lopinavir/ritonavir arm was later dropped in Version 3.0, and only Version 2.0 women who received efavirenz or raltegravir were included in the study analyses. Therefore, because no women included in the study analyses received lopinavir/ritonavir, this outcome measure was not analyzed.
Time Frame: Measured on or after delivery up to participants' last postpartum study visit (approximately 26 weeks after delivery)
Population: Because the study arm that was associated with this outcome measure was dropped, no women were assessed for this outcome.
Arm/Group | Arm A (Women) | Arm B (Women)
Number analyzed (Participants) | 0 | 0

11. Secondary Outcome: Proportion of Deliveries That Had an Outcome of a Stillbirth/Fetal Demise.
Description: The unit of analysis was the mother-infant set. All sets where the woman received at least one dose of study treatment and remained on study through delivery were eligible. In the case of twins, the worst outcome (i.e. a stillbirth) was used.
Time Frame: Measured at delivery (approximately 36 to 40 weeks gestation)
Population: Fourteen women (8 in Arm A and 6 in Arm B) were off-study prior to delivery (including the 5 women in Arm A who never initiated study treatment).
Measure: Number; unit: Proportion
Arm/Group | Arm A (Women) | Arm B (Women)
Number analyzed (Participants) | 194 | 200
Proportion | .005 | .015
Statistical Analysis 1: Comparison: Arm A (Women) vs Arm B (Women); Test type: Superiority; p = 0.623, Fisher Exact

12. Secondary Outcome: Proportion of Deliveries That Were Premature (Less Than 37 Weeks Gestation)
Description: The unit of analysis for this outcome measure was the mother-infant set. A mother-infant set was counted as having a premature delivery if any infant in the mother-infant set was delivered prior to 37 weeks gestation (i.e. in the case of twins, if either of the twins was delivered prior to 37 weeks gestation then this set would count as one premature delivery outcome).
  All mother-infant sets that delivered at least one live birth on study were eligible for this outcome.
Time Frame: Measured at delivery (within 72 hours).
Population: There were 393 live-birth infants on study. There were three sets of twins, leaving 390 mother-infant sets that delivered at least one live birth on study. Five sets (three EFV and two RAL) did not have gestational age at delivery recorded and were excluded, leaving 385 sets included in this outcome.
Measure: Number; unit: Proportion
Arm/Group | Arm A (Women) | Arm B (Women)
Number analyzed (Participants) | 190 | 195
Proportion | .105 | .123
Statistical Analysis 1: Comparison: Arm A (Women) vs Arm B (Women); Test type: Superiority; p = .63, Fisher Exact

13. Secondary Outcome: Proportion of Deliveries That Were Extremely Premature (Less Than 34 Weeks Gestation).
Description: The unit of analysis for this outcome measure was the mother-infant set. A mother-infant set was counted as having an extremely premature delivery if any infant in the mother-infant set was delivered prior to 34 weeks gestation (i.e. in the case of twins, if either of the twins was delivered prior to 34 weeks gestation then this set would count as one extremely premature delivery outcome).
  Only women who enrolled prior to 34 weeks gestation were included in this analysis. Those that enrolled from 34 to less than 37 weeks gestation were excluded because they were already past the gestational age where this outcome could have occurred at entry.
Time Frame: At delivery (within 72 hours).
Population: There were 393 live-birth infants on study. There were three sets of twins, leaving 390 mother-infant sets that delivered at least one live birth on study. Among these, five were missing gestational age at delivery (three EFV and two RAL sets) and 45 were enrolled from 34 to less than 37 weeks gestation and excluded, leaving 340 evaluable sets.
Measure: Number; unit: Proportion
Arm/Group | Arm A (Women) | Arm B (Women)
Number analyzed (Participants) | 169 | 171
Proportion | .036 | .023
Statistical Analysis 1: Comparison: Arm A (Women) vs Arm B (Women); Test type: Superiority; p = .54, Fisher Exact

14. Secondary Outcome: Proportion of Deliveries With a Low Birth Weight (Less Than 2,500 Grams)
Description: The unit of analysis was the mother-infant pair or set; in the case of multiple gestation, the worst outcome was considered in analysis (e.g. if two twins were delivered to one mother, one at 2,000 grams and one at 3,000 grams, this mother-infant set would count as one instance of low birth weight in analysis because at least one of the infants had the outcome).
Time Frame: Measured within 72 hours after delivery
Population: All women who delivered at least one live-birth infant on-study were included in this analysis. Although 393 live-born infants were delivered, there were three sets of twins. Therefore, 390 mother-infant pairs were included in this analysis.
Measure: Number; unit: Proportion
Arm/Group | Arm A (Women) | Arm B (Women)
Number analyzed (Participants) | 193 | 197
Proportion | .124 | .127
Statistical Analysis 1: Comparison: Arm A (Women) vs Arm B (Women); Test type: Superiority; p > 0.99, Fisher Exact

15. Secondary Outcome: Proportion of Deliveries With an Extremely Low Birth Weight (<1,500 Grams).
Description: The unit of analysis was the mother-infant pair or set; in the case of multiple gestation, the worst outcome was considered in analysis (e.g. if two twins were delivered to one mother, one at 2,000 grams and one at 1,000 grams, this mother-infant set would count as one instance of extremely low birth weight in analysis because at least one of the infants had the outcome).
Time Frame: Measured within 72 hours after delivery
Population: as for outcome 14
Measure: Number; unit: Proportion
Arm/Group | Arm A (Women) | Arm B (Women)
Number analyzed (Participants) | 193 | 197
Proportion | .000 | .005
Statistical Analysis 1: Comparison: Arm A (Women) vs Arm B (Women); Test type: Superiority; p > 0.99, Fisher Exact

16. Secondary Outcome: Infant HIV Infection Status (Per International Maternal Pediatric Adolescent AIDS Clinical Trials Group [IMPAACT] Definitions)
Description: Infants were considered infected if they had both a positive HIV nucleic acid test and a subsequent confirmatory test on a different sample. Uninfected infants were those that had no positive test results and negative test results obtained at two or more of the following visits: Week 6, Week 16, and/or Week 24 postpartum.
Time Frame: Measured from birth through infants' last study visit at Week 24
Population: Infants who had no positive test result, but did not have negative results at at least two of Week 6, 16, and/or 24 postpartum visits were not eligible for this analysis. All infants who had at least one positive test also had a positive confirmation test, and are included in this outcome.
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A (Infants) | Arm B (Infants)
Number analyzed (Participants) | 184 | 190
Participants
  HIV-infected | 6 | 1
  HIV-uninfected | 178 | 189
Statistical Analysis 1: Comparison: Arm A (Infants) vs Arm B (Infants); The proportion of HIV-infected infants among those who had a determinable HIV-infection status was compared between arms; Test type: Superiority; p = 0.064, Fisher Exact

17. Secondary Outcome: Proportion of HIV-infected Infants With Genotypic Resistance to Study Drugs
Description: Genotypic resistance to each class of study drug (reverse transcriptase inhibitors and integrase inhibitors) was assessed separately among HIV infected infants.
Time Frame: Measured on or after confirmation of HIV-infection up to the infants' last study visit at Week 24
Population: One infant in the efavirenz arm did not have a specimen collected with sufficient viral load to perform consensus sequencing. All other infected infants had genotypic resistance results for both classes of study drug.
Measure: Number; unit: Proportion
Arm/Group | Arm A (Infants) | Arm B (Infants)
Number analyzed (Participants) | 5 | 1
Proportion
  Reverse transcriptase resistance | .20 | .00
  Integrase resistance | .00 | .00

18. Secondary Outcome: Proportion of Women With HIV-1 Drug Resistance Mutations at Screening, 2-4 Weeks Postpartum in Women Who Stopped Antiretroviral Therapy, and at the Time of Inadequate Virologic Response Using Standard and Ultrasensitive Methods.
Description: Consensus sequencing was performed on a sample from screening. Women were evaluated for integrase and reverse transcriptase resistance mutations separately.
  Additionally, consensus sequencing was performed among women who had an inadequate virologic response (defined in the protocol) on a sample taken at that time of inadequate virologic response.
  Genotypic resistance among women who stopped antiretroviral therapy was not assessed. Because World Health Organization guidelines have been updated to indicate all people living with HIV should remain on antiretroviral therapy, even postpartum women, no women stopped antiretroviral therapy after delivery. Therefore, this aspect of the outcome measure is no longer relevant and was not assessed.
Time Frame: Measured at screening and at the time of inadequate virologic response (from Week 2 antepartum through participants' last study visit 24 weeks after delivery).
Population: Women were excluded if they had indeterminate or unknown resistance results for that class of antiretroviral study drug.
Measure: Number; unit: Proportion
Arm/Group | Arm A (Women) | Arm B (Women)
Number analyzed (Participants) | 190 | 197
Proportion
  Reverse transcriptase resistance at screening: number analyzed (Participants) | 187 | 197
  Reverse transcriptase resistance at screening | .07 | .11
  Integrase resistance at screening: number analyzed (Participants) | 190 | 192
  Integrase resistance at screening | .00 | .00
  Reverse transcriptase resistance at viral failure: number analyzed (Participants) | 5 | 10
  Reverse transcriptase resistance at viral failure | .60 | .30
  Integrase resistance at viral failure: number analyzed (Participants) | 0 | 10
  Integrase resistance at viral failure |  | .00

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from entry (20-36 weeks gestation) through delivery for women. Additionally, both women and infants had adverse event data collected from delivery through their final study visit which was scheduled to occur at Week 24 postpartum.
Description: Serious adverse events and deaths were reported among all women and live-birth infants. Only women who received at least one dose of study drug (and their infants) were included in the assessment of "other" events, which included grade 3 or higher signs/symptoms, laboratory events, and diagnoses that occurred in at least 5 percent of women (or infants) in at least one arm.
  The DAIDS AE Grading Table (V2.0) and EAE Manual (V2.0) were used.
Arm/Group | Arm A (Women) | Arm B (Women) | Arm A (Infants) | Arm B (Infants)
All-Cause Mortality (participants affected / at risk) | 0/197 | 1/206 | 1/194 | 1/199
Serious Adverse Events (participants affected / at risk) | 34/202 | 34/206 | 31/194 | 50/199
Other Adverse Events (participants affected / at risk) | 20/197 | 24/206 | 20/194 | 15/199
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (Women) (N=202) | Arm B (Women) (N=206) | Arm A (Infants) (N=194) | Arm B (Infants) (N=199)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ABO incompatibility (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Abortion threatened (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Alanine aminotransferase increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Anaemia (Blood and lymphatic system disorders) | 2 (2) | 0 (0) | 3 (3) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Atrial septal defect (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 4 (4)
Bilirubin conjugated increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Blood bilirubin increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cardiac murmer (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital cytomegalovirus infection (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital pneumonia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Congenital syphilis (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 12 (12) | 12 (12)
Congenital toxoplasmosis (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erysipelas (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foetal distress syndrome (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 5 (5) | 0 (0) | 0 (0)
Gastroenteritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Genitalia external ambiguous (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Haemoglobin decreased (Investigations) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
Hepatic rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatotoxicity (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Herpes simplex encephalitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydrocephalus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hyperbilirubinaemia neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 1 (1) | 5 (5) | 0 (0) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hypospadias (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neonatal asphyxia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Neonatal respiratory distress (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neonatal respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) | 0 (0) | 0 (0)
Overdose (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pelvis abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Polyhydramnios (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postpartum haemorrhage (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Pre-eclampsia (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 3 (3) | 0 (0) | 0 (0)
Premature baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 3 (3) | 4 (4)
Premature labor (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Puerperal pyrexia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pulmonary artery stenosis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary valve stenosis (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyloric stenosis (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
Respiratory syncytial virus bronchiolitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Sepsis neonatal (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 4 (4)
Sudden infant death syndrome (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Suicidal ideation (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Talipes (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Transient tachypnoea of the newborn (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Tricuspid valve incompetance (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Umbilical cord around neck (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Umbilical hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ankyloglossia (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
Single umbilical artery (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Infection prophylaxis (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Macrocephaly (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Necrotising colitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foetal death (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Bicytopenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hepatic enzyme increased (Investigations) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Foetal malformation (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pneumonia bacterial (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Pyelocaliectasis (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Extrapulmonary tuberculosis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Low birth weight baby (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hypoxic-ischaemic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Foetal growth restriction (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Gestational hypertension (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 2 (2) | 0 (0) | 0 (0)
Congenital skin dimples (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Escherichia pyelonephritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Meconium aspiration syndrome (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A (Women) (N=197) | Arm B (Women) (N=206) | Arm A (Infants) (N=194) | Arm B (Infants) (N=199)
Haemoglobin decreased (Investigations) | 20 | 24 | 10 | 3
Congenital syphilis (Congenital, familial and genetic disorders) | 0 | 0 | 12 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-02-28): https://cdn.clinicaltrials.gov/large-docs/05/NCT01618305/SAP_000.pdf
  • Study Protocol (2015-04-02): https://cdn.clinicaltrials.gov/large-docs/05/NCT01618305/Prot_001.pdf